CLINICAL TRIAL: NCT04792450
Title: Thales Thermography Triage (3T) - Pilot Project: Developing a Thermal Camera That Accurately Records Participants' Temperature From Images of Their Face
Brief Title: Thales Thermography Triage (3T) - Pilot Project
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: NHS Greater Clyde and Glasgow (Other)
Collaborators: Thales Group (Unknown)
Responsible Party: Principal Investigator, David Lowe, Dr David J Lowe, NHS Greater Clyde and Glasgow
Other Study IDs: 287901
Record Dates: First submitted 2020-09-25; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Fever
MeSH Terms: conditions — Fever | interventions — Thermography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ED Patients: Patients presenting in Emergency Department
  Interventions: Device: Thermography; Device: Tympanic Thermometer; Device: Forehead Thermometer; Device: 62 Max + Infra-red thermometer
- ED Staff: Staff working within the Emergency Department
  Interventions: Device: Thermography; Device: Tympanic Thermometer; Device: Forehead Thermometer; Device: 62 Max + Infra-red thermometer

INTERVENTIONS:
Device: Thermography — Measure Temperature using Thermal Camera
Device: Tympanic Thermometer — Measure Temperature using Tympanic Thermometer
Device: Forehead Thermometer — Measure Temperature using Forehead Temperature
Device: 62 Max + Infra-red thermometer — Measure Temperature using 62 Max + Infra-red thermometer

SUMMARY:
COVID Related Study.

This study will compare the Thales High Temperature Detection (HTD) system with the two routinely used temperature measurement systems (tympanic and forehead) in patients and staff in the Emergency Department.

The aims of the study are:

* To determine the diagnostic accuracy of HTD for the measurement of fever, using an equivalence comparison with the maximum temperature recorded with two routinely used temperature measurements (tympanic and forehead), margin ±0.2°C.
* To determine if skin tone is an independent confounding factor in the measurement of fever using HTD
* To establish performance of internal calibration of Thales device
* To power for a definitive Clinical Investigation to determine clinical efficacy and safety cut off with HTD If results are encouraging the aim would then be to undertake a clinical investigation in order to get CE marking for use in a clinical setting.

DETAILED DESCRIPTION:
In the fifty years since the emergence of thermal imaging technology, Thales in Glasgow has built up a world leading capability in the design, manufacture and supply of Thermal Imaging cameras. In addition to the cameras, Thales in Glasgow has a particular expertise in developing image processing algorithms (conventional and artificial intelligence based) to allow the cameras to perform critical user tasks beyond mere imaging.

COVID-19 [SARS-COV-2] has placed a huge challenge on the world. In response to the crisis, Thales is engaged in a number of initiatives, including one aimed at the possible application of thermal imaging cameras to detect people with a fever and hence those who may be suffering from COVID-19.Fever is a key symptom of covid-19. One of the major limitations of existing systems is thermographic accuracy. Most current thermographic camera systems offer an accuracy of ± 0.5°C. This can be reduced to ±0.3°C with the inclusion of a "Black Body" calibration source, although this limits the portability of the system. Using their unique knowledge and expertise in high resolution and precision thermal imaging and thermal image processing, Thales aims to develop a fever screening system with an accuracy of ± 0.1°C to enable more effective identification and triage of people with fever.

What Thales lacks is real world thermal images of patients suffering fever and access to clinicians who can advise on the medical aspects of the work. This research would fill these two voids.

In a pilot study conducted in the Emergency Department, Queen Elizabeth University Hospital (20/NS/0064), the Thales High Temperature Detection (HTD) system was found to be more accurate than a tympanic thermometer which captures Infrared radiation emitted by the tympanic membrane in the ear or forehead thermometer. Tympanic temperature measurements are typically used in the hospital setting in Scotland whereas forehead IR measurement is common in transportation and workplace settings.

The HTD has been redesigned in response to three key findings from the pilot study:

* The relative temperature of some facial features correlated more strongly with tympanic temperature than others.
* Having an external Black Body (BB) calibration source in the scene at all times was impractical in a clinical environment
* Camera systems require to be compact and portable to be useful to clinical staff.

As a result, the HTD is now significantly reduced in size, including peripheral devices. A novel calibration solution has been designed (and patented) that not only removes the need for the black body source but allows for a more accurate temperature evaluation. In addition, facial feature detection has been integrated into the software to allow it to automatically locate the patient's head and in the near future, automatically determine the temperatures of individual facial features. This development will capture facial feature detection - not facial recognition.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 16 years old with no upper age limit
* Patients able to read and understand English
* Patients able to give informed consent
* Patients being triaged through ED for any complaint, not necessarily COVID-19 QEUH ED staff

Exclusion Criteria:

* Patients not meeting the inclusion criteria
* Patients who do not have capacity to consent
* Patients attending ED who are fast-tracked without triage

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients attending Queen Elizabeth University Hospital Emergency Department requiring triage. All staff members working within Queen Elizabeth University Hospital Emergency Department.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2020-12-15 (Actual); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
To determine the diagnostic accuracy of HTD for the measurement of fever, using an equivalence comparison with the maximum temperature recorded with two routinely used temperature measurements (tympanic and forehead), margin ±0.2°C. | First 4 hours of hospitalisation.
  Measurement of temperature in celsius

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Elizabeth University Hospital, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2020-09-09): https://cdn.clinicaltrials.gov/large-docs/50/NCT04792450/Prot_000.pdf